CLINICAL TRIAL: NCT00738309
Title: Prospective Study of Scheuermann's Kyphosis
Acronym: PSK
Status: Completed | Type: Observational
Sponsor: Setting Scoliosis Straight Foundation (Other)
Collaborators: DePuy Spine (Industry)
Responsible Party: Sponsor
Other Study IDs: 2006HSGDEF13
Record Dates: First submitted 2008-08-18; First posted 2008-08-20 (Estimated); Last update posted 2016-04-19 (Estimated); Status verified 2016-04

CONDITIONS: Scheuermann's Kyphosis
Keywords: Treatment Outcomes; Spinal Deformity; Scheuermann's Kyphosis
MeSH Terms: conditions — Scheuermann Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Operative: Diagnosis of classical Scheuermann's Kyphosis (3 successive vertebrae wedged 5 degrees or more, +/- end plate deformities) or idiopathic structural Kyphosis (rigid structural kyphosis without classic Scheuermann's Kyphosis findings) for which surgical treatment is recommended to prevent progression of the curvature or to correct trunk deformity (unacceptable cosmesis).
- Non-operative: Diagnosis of classical Scheuermann's Kyphosis (3 successive vertebrae wedged 5 degrees or more, +/- end plate deformities) or idiopathic structural Kyphosis (rigid structural kyphosis without classic Scheuermann's Kyphosis findings) for which surgical treatment was not undertaken.

SUMMARY:
The purpose of this study to determine the radiographic and clinical outcomes of spinal deformity surgical treatment in patients with Scheuermann's Kyphosis.

ELIGIBILITY:
Inclusion Criteria:

* Patient age < 21 years
* Male or female
* Diagnosis of classical Scheuermann's Kyphosis (3 successive vertebrae wedged 5 degrees or more, +/- end plate deformities) or idiopathic structural Kyphosis (rigid structural kyphosis without classic Scheuermann's Kyphosis findings).
* for which surgical treatment is recommended to prevent progression of the curvature or to correct trunk deformity (unacceptable cosmesis) - any deformity magnitude.

OR

* for which surgical treatment is not being undertaken (and alternate treatment, i.e. bracing, or observation) is being pursued for any curve magnitude of clinical concerns of Scheuermann's Kyphosis.
* Inclusion Criteria for Anterior Release (for those surgeons performing anterior release surgery): Deformity magnitude = any degree and any other criteria defined by the individual surgeon.
* Posterior disc herniation is not an exclusion criteria from being in the study, only from being in the Posterior surgery group - these patients will be defaulted to Ant/Post Surgery.
* Only patients that have had a pre-op MRI performed as a part of their routine care, should be included in this study.

Exclusion Criteria:

* Previous operated Kyphosis, Scoliosis or Spondylolisthesis
* Neuromuscular co-morbidity
* Post laminectomy kyphosis

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients who present to the investigator's clinic, who meet the inclusion criteria will be offered enrollment in the study.
Sampling Method: Non-Probability Sample
Enrollment: 147 (Actual)
Dates: Start 2006-05; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
radiographic outcomes | 2 years

SECONDARY OUTCOMES:
Clinical outcomes | 2 years
Health related quality of life outcomes | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Baron Lonner, MD, Principal Investigator — Scoliosis Associates - New York, NY; Peter Newton, MD, Study Director — Rady Children's Hospital, San Diego; Michelle C Marks, PT, MA, Study Chair — Harms Study Group
Locations (9):
- United States (8):
  - UC Davis, Sacramento, California
  - Rady Children's Hospital, San Diego, California
  - A.I. DePont Hospital for Children, Wilmington, Delaware
  - Miami Children's Hospital, Miami, Florida
  - John's Hopkins Medical Institute, Baltimore, Maryland
  - University Physicians, Camden, New Jersey
  - Cincinnati Children's Hospital, Cincinnati, OH, Cincinnati, Ohio
  - Shriners Hospital for Children, Philadelphia, Pennsylvania
- Rehabilitationskrankenhaus Lagensteinbach, Lagensteinbach, Karlsbad, Germany